CLINICAL TRIAL: NCT01911195
Title: Reconstructing Consciousness and Cognition
Acronym: RCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Pennsylvania (Other); Washington University School of Medicine (Other); James S McDonnell Foundation (Other)
Responsible Party: Principal Investigator, George Mashour, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: McDonnell RCC
Record Dates: First submitted 2013-07-21; First posted 2013-07-30 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: General anesthesia; cognition; consciousness
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Cognitive Testing (Active Comparator): Control arm will receive cognitive testing only without undergoing general anesthesia
  Interventions: Other: Control Group: Cognitive Testing
- ISOFLURANE- Experimental Arm (Experimental): Experimental arm will receive cognitive testing before and after general anesthesia
  Interventions: Drug: ISOFLURANE- Experimental Arm

INTERVENTIONS:
Drug: ISOFLURANE- Experimental Arm — The experimental group will be given the anesthetic isoflurane for three hours, and will undergo cognitive tests immediately following emergence from general anesthesia while connected to an EEG machine.
  Arms: ISOFLURANE- Experimental Arm
Other: Control Group: Cognitive Testing — The control group will undergo cognitive testing while connected to an EEG machine following a comparable rest period, but will not receive general anesthesia.
  Arms: Control Group: Cognitive Testing

SUMMARY:
Currently it is unknown how the human brain reorganizes its network organization to generate conscious experience and cognitive activity after a period of unconsciousness. Therefore, the purpose of this study is to assess how cognitive activity is reconstructed after general anesthesia. The investigators hypothesize that the brain's transition from unconsciousness to consciousness and full cognition is a complex process that occurs over an extended period of time. Specifically, the investigators hypothesize the following order of cognitive reconstitution: responsiveness to command, attention, complex scanning and visual tracking, working memory, and executive function.

Volunteers will be healthy participants who are anesthetized with commonly used anesthetic drugs as well as a non-anesthetized group to control for circadian influences. A total of 60 subjects will be recruited for this study. All subjects (male and female) will perform basic tests for cognition on a laptop computer at 30-minute intervals during this study. The testing battery to be administered was assembled to assess multiple cognitive functions in order to determine whether and how cognitive processes return to baseline function. Electroencephalogram (measuring brain electrical activity) data will be monitored and recorded during both anesthesia and cognitive testing, for subsequent analysis.

This study is significant because it could lead to a better understanding of the neural correlates of human consciousness, as well as normal and abnormal conscious state transitions (including barriers to such transitions).

ELIGIBILITY:
Inclusion Criteria:

* Healthy 20-40 year old volunteers,
* American Society of Anesthesiologists Physical Status I or II (i.e., healthy),
* Body mass index < 30 kg/m2,
* Easily visualized uvula,
* With anticipated equal recruitment of males and females.

Exclusion Criteria:

* Physical signs suggestive of difficult airway (e.g., mouth opening <3cm, short distance between the chin and neck, poor mandibular subluxation, thick neck),
* History of obstructive sleep apnea,
* Reactive airway disease,
* Neuropsychiatric disorders,
* History or current use of psychotropic medications,
* Current tobacco and alcohol use,
* History of hypertension or current medication for blood pressure control, cardiovascular disease or arrhythmias,
* Positive urine toxicology screen,
* History of reflux,
* Pregnancy,
* Family history of problems with anesthesia (including but not limited to malignant hyperthermia),
* Sleep disorders,
* History of postoperative nausea/vomiting or motion sickness,
* Allergy to eggs, egg products or soy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-02-09 (Actual); Study Completion 2015-02-09 (Actual)

PRIMARY OUTCOMES:
Neurocognitive scores | Three hours following emergence from general anesthesia
  Neurocognitive battery performed on computer

SECONDARY OUTCOMES:
Brain network connectivity | Three hours following emergence from general anesthesia
  Functional brain networks will be reconstructed from EEG data.

CONTACTS AND LOCATIONS:
Overall Officials: George A Mashour, MD, PhD, Principal Investigator — University of Michigan; Michael Avidan, MBBCh, Principal Investigator — Washington University School of Medicine; Max Kelz, MD, PhD, Principal Investigator — University of Pennsylvania; Mathias Basner, MD, PhD, MSc, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Mashour GA, Palanca BJ, Basner M, Li D, Wang W, Blain-Moraes S, Lin N, Maier K, Muench M, Tarnal V, Vanini G, Ochroch EA, Hogg R, Schwartz M, Maybrier H, Hardie R, Janke E, Golmirzaie G, Picton P, McKinstry-Wu AR, Avidan MS, Kelz MB. Recovery of consciousness and cognition after general anesthesia in humans. Elife. 2021 May 10;10:e59525. doi: 10.7554/eLife.59525. PMID 33970101
- [Derived] Labonte AK, Kafashan M, Huels ER, Blain-Moraes S, Basner M, Kelz MB, Mashour GA, Avidan MS, Palanca BJA; ReCCognition Study Group. The posterior dominant rhythm: an electroencephalographic biomarker for cognitive recovery after general anaesthesia. Br J Anaesth. 2023 Feb;130(2):e233-e242. doi: 10.1016/j.bja.2022.01.019. Epub 2022 Feb 17. PMID 35183346